CLINICAL TRIAL: NCT02391571
Title: A Randomized, Double-Blind, Multiple-Dose, Parallel Group Study to Evaluate the Potential of Withdrawal Effects Following Administration of Oxycodone/Naltrexone Capsules and Oxycodone in Methadone-Maintained Opioid-Dependent Subjects
Brief Title: A Study to Evaluate Withdrawal Effects Following Dosing of Oxycodone/Naltrexone in Methadone-Maintained Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Elite Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: ELI-004-2015
Record Dates: First submitted 2015-02-17; First posted 2015-03-18 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Withdrawal Symptoms
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Oxycodone; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxycodone/Naltrexone (Experimental): Oxycodone/Naltrexone Capsules (over-encapsulated), on days 6-10, every 6 hours (at 09:00, 15:00, 21:00)
  Interventions: Drug: Oxycodone/Naltrexone Capsules
- Oxycodone (Active Comparator): Oxycodone Tablets (Over-encapsulated), on Days 6-10, every 6 hours (at 09:00, 15:00, 21:00)
  Interventions: Drug: Oxycodone
- Placebo Lead-In (Other): Placebo Lead-In: Placebo Capsules (matching to Active and Experimental) on days 4-5, every 6 hours (at 09:00, 15:00, 21:00)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone/Naltrexone Capsules — Oxycodone/Naltrexone to be taken with stable dose of Methadone
  Arms: Oxycodone/Naltrexone
Drug: Oxycodone — Oxycodone to be taken with stable dose of Methadone
  Arms: Oxycodone
Drug: Placebo — 2 day placebo run in prior to test and active drug phase of study
  Arms: Placebo Lead-In

SUMMARY:
This single-center study is a randomized, double-blind, active-controlled, multiple-dose, parallel group study to evaluate the potential withdrawal effects, safety and tolerability, and pharmacokinetic and pharmacodynamic effects of multiple doses of oral intact Oxycodone/Naltrexone capsules compared to oxycodone in methadone-maintained opioid-dependent subjects. The study will consist of a Screening Phase, an inpatient Treatment Phase (including a methadone stabilization period, a placebo administration period, a treatment administration period and a safety/washout period), and a Follow-up Phase.

DETAILED DESCRIPTION:
Approximately 34 methadone-maintained opioid-dependent subjects will be enrolled in the study. All subjects will be admitted to the clinical study unit (CSU; Visit 2) for a 15-day (with 14 overnight stays) inpatient Treatment Phase visit. Subjects will first undergo a 3-day methadone stabilization period (Days 1 to 3) in which all subjects' methadone administration time will be gradually shifted to the time of dosing that will be used throughout the Treatment Phase (approximately 8 am daily). Following the methadone dosing-time stabilization period, subjects will begin a 2-day oxycodone placebo administration period. On Day 4 and Day 5, all subjects will receive a total of 3 oxycodone placebo doses, separated by 6 hours each, starting from approximately one hour following methadone dose administration. Placebo will be administered in a single-blind manner. Starting on Day 6, subjects will be randomized in a 2:1 (Oxycodone/Naltrexone or Oxycodone) fashion to receive one of the following treatments in a double-blinded manner:

* Oxycodone/Naltrexone, multiple oral daily dosing for 5 days
* Oxycodone, multiple oral daily dosing for 5 days Subjects will receive one of the above-listed treatments three times daily, beginning approximately 1 hour following methadone dosing and every 6 hours until 3 doses have been administered. Subjects will be dosed in this manner for 5 consecutive days (Days 6 to 10). All subjects will remain confined in the CSU for 4 days after the first of three doses of study drug is administered on Day 10 for the safety/washout period, during which they will continue to be assessed and monitored for withdrawal effects. Subjects will be discharged approximately 96 hours after the first dose of study drug (oxycodone/naltrexone or oxycodone) administered on the morning of Day 10, if medically acceptable according to the investigator or designee. All subjects will receive daily phone calls until the Follow-up Phase during which subjects will be asked about the presence of withdrawal symptoms and any other adverse events (AEs).

On Days 4 to 9, safety, withdrawal, pharmacokinetic and pharmacodynamic assessments will be performed up to 13 hours after the first of the three daily study drug doses is administered. Following Day 10 study drug administration, assessments will be completed until 96 hours after the first of the three daily study drug doses is administered on the morning of Day 10.

The Follow-up Phase will be conducted approximately 10 to 14 days after the last drug administration on Day 10 or after early withdrawal from the study and will include standard safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects 18 to 55 years of age, inclusive.
2. Body mass index (BMI) within the range of 18.0 to 35.0 kg/m2, inclusive, and a minimum weight of 50.0 kg.
3. Maintained on a stable methadone regimen. Subjects must be receiving a methadone dose of 50 to 150 mg/day at Screening, with dosage variation ≤20% for at least 14 days prior to the Screening visit and who are willing to remain on their dose at Screening and for the duration of the study.
4. The study volunteer has been previously exposed to opioids while on methadone maintenance without relapse occurring, or in the opinion of the methadone maintenance program Director or Physician, is not at undue risk of relapse from participation in the clinical study.

Exclusion Criteria:

1. History or presence of clinically significant abnormality as assessed by physical examination, medical history, 12-lead ECG, vital signs, or laboratory values, which in the opinion of the investigator would jeopardize the safety of the subject or the validity of the study results.
2. Clinically significant infection/injury/illness within 1 month prior to Screening.
3. Has been diagnosed with cancer within 5 years prior to screening (excluding squamous or basal cell carcinoma of the skin), or has an active malignancy of any type (including squamous or basal cell carcinoma of the skin).
4. History of major mental illness that in the opinion of the investigator may affect the ability of the subject to participate in the study. Institutionalized subjects will not be eligible for participation.
5. Documented history of a medical condition that, in the opinion of the investigator, would compromise the subject's ability to swallow, absorb, metabolize, or excrete test product, including (but not limited to) intractable nausea and/or vomiting and/or severe gastrointestinal narrowing (pathologic or iatrogenic).
6. Documented history of, or currently active, seizure disorder or history of clinically significant head injury or syncope of unknown origin.
7. History of severe allergic reaction (including anaphylaxis) to any substance, or previous status asthmaticus, or food allergies/intolerances/restrictions, or special dietary needs which, in the judgment of the investigator, contraindicates the subject's participation in the study.
8. History of allergy or hypersensitivity to oxycodone or related drugs (e.g., other opioids) or naltrexone or related drugs (e.g., other antagonists).
9. 13. An employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member defined as a spouse, parent, child or sibling, whether biological or legally adopted.
10. A subject who, in the opinion of the investigator or designee, is considered unsuitable or unlikely to comply with the study protocol for any reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Primary: Onset of Withdrawal measured by Subjective Opioid Withdrawal Scale(SOWS) | up to 10 days
  To assess the withdrawal effects of intact Oxycodone/Naltrexone following multiple dose administration compared to Oxycodone in methadone-maintained, opioid-dependent subjects (all subjects enrolled in the study N=34) over time using Subjective Opioid Withdrawal Scale(SOWS), a set of 16 questions scored on a scale of 0-4 (not at all to extremely) according to how the subject feels at that moment to the questions asked about withdrawal symptoms. The questions are asked during the placebo period 9 times daily , and daily during treatment administration 9 times a day.
Primary: Onset of Withdrawal measured by Clinician-Rated Opioid Withdrawal Scale (COWS) | up to 10 days
  To assess the withdrawal effects of intact Oxycodone/Naltrexone following multiple dose administration compared to Oxycodone in methadone-maintained, opioid-dependent subjects (all subjects enrolled in the study N=34) over time using Clinician-Rated Opioid Withdrawal Scale (COWS), a set of 11 questions scored by a trained clinician that best describes the subject's signs or symptoms of withdrawal at that time. Each are rated on the apparent relationship to opiate withdrawal. These are assessed during the placebo period 9 times daily , and daily during treatment administration 9 times a day. A total score is tallied that determines mild, moderate, moderately severe or severe withdrawal.

SECONDARY OUTCOMES:
Secondary: Pharmacokinetic Profile of Naltrexone and 6β-Naltrexol in Subjects receiving Oxycodone/Naltrexone | up to 14 days
  To investigate the multiple dose pharmacokinetics of naltrexone, and 6β-naltrexol following repeated daily administration of Oxycodone/Naltrexone in methadone-maintained opioid dependent subjects. All subjects enrolled will have 3 PK samples taken during the placebo period and 3-13 samples taken during days 6-10 of the study. Samples will also be taken during the wash-out period, 2 on Day 11, then daily through Day 14. T max, Cmax AUC Ctrough and apparent first-order terminal elimination half-life will be calculated as part of the PK profile.
Secondary: Subjective Pharmacodynamic Effects through the use of Visual Analog Scales (VAS) | up to 14 days
  To explore the pharmacodynamic effects of Oxycodone/Naltrexone following multiple dose administration compared to Oxycodone in methadone maintained opioid-dependent subjects through the use of Visual Analog Scales (VAS) to rate Bad Effects, Feeling Sick and Any Effects at the moment of the scale being administered, with 0 mm being "Not At All" and 100 mm being "Extremely". These are administered during the placebo period 9 times daily , and daily during treatment administration 9 times a day. Also, the measurement will be taken during the wash-out period daily. All enrolled subjects will have the VAS measurements administered.
Secondary: Objective Pharmacodynamic Effects through the use of Pupillometry measurements | up to 14 days
  To explore the physiological effects of Oxycodone/Naltrexone following multiple dose administration compared to Oxycodone in methadone maintained opioid-dependent subjects through the use of Pupillometry measurements. An electronic pupillometry will be used, and every effort will be made to use the same eye for each measurement. Measurements will be taken during the placebo period 9 times daily , and daily during treatment administration 9 times a day. Also, the measurement will be taken daily during the wash-out period. All enrolled subjects will have the pupillometry measurements taken.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Vince and Associates
Locations (1):
- Vince and Associates, Overland Park, Kansas, United States